CLINICAL TRIAL: NCT04173416
Title: The Youth Opioid Recovery Support (YORS) Intervention: An Assertive Community Treatment Model for Improving Medication Adherence in Young Adults With Opioid Use Disorder
Brief Title: The Youth Opioid Recovery Support (YORS) Intervention
Acronym: YORS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Potomac Health Foundations (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Friends Research Institute, Inc. (Other); National Center for Complementary and Integrative Health (NCCIH) (NIH); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R61AT010614 (NIH); R61AT010614 (NIH)
Record Dates: First submitted 2019-11-20; First posted 2019-11-22 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Opioid-use Disorder; Medication Adherence
MeSH Terms: conditions — Opioid-Related Disorders; Medication Adherence

STUDY DESIGN:
Intervention Model Description: Phase 1 of the study (years 1-2) will include a single group, open-label, intervention only arm. After iterative cycles of testing and refinement, we will proceed with a parallel group RCT in Phase 2 of the study (years 3-5).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Youth Opioid Recovery Support (YORS) (Experimental): The Youth Opioid Recovery Support (YORS) model is an innovative wrap-around approach that attempts to address barriers to treatment engagement in this vulnerable young adult population, especially difficulties with medication adherence. Its components include: (1) Home delivery of extended release naltrexone (XR-NTX) for OUD; (2) Engagement of families in collaborative treatment planning and monitoring focusing on medication adherence; (3) Assertive outreach from the treatment team including actively tracking and communicating with youth and families by text messaging and social media to promote engagement and adherence; and (4) Contingency management to provide incentives for medication adherence.
  The specific components of YORS will be refined and adapted based on feedback from interviews and focus groups with various stakeholders. However, the basic framework outlined above is expected to persists.
  Interventions: Behavioral: Youth Opioid Recovery Support (YORS)
- Treatment As Usual (No Intervention): TAU will contain patients who will be receiving treatment for opioid use disorder through their usual venues without the family engagement, assertive outreach, contingency management, and home delivery of medication. This often includes a referral and warm hand off to intensive outpatient SUD services and/or mental health care.

INTERVENTIONS:
Behavioral: Youth Opioid Recovery Support (YORS) — The Youth Opioid Recovery Support (YORS) model is an innovative wrap-around approach that attempts to address barriers to treatment engagement in this vulnerable young adult population, especially difficulties with medication adherence. Its components include: (1) Home delivery of extended release naltrexone (XR-NTX) for OUD; (2) Engagement of families in collaborative treatment planning and monitoring focusing on medication adherence; (3) Assertive outreach from the treatment team including actively tracking and communicating with youth and families by text messaging and social media to promote engagement and adherence; and (4) Contingency management to provide incentives for medication adherence.
  Arms: Youth Opioid Recovery Support (YORS)

SUMMARY:
Youth are disproportionately affected by the current opioid crisis with catastrophic consequences, and young adults with opioid use disorder (OUD) often struggle with adherence to relapse prevention medications. The Youth Opioid Recovery Support (YORS) model is a promising, innovative, wrap-around approach that addresses barriers to medication adherence and treatment engagement in an effort to improve public health outcomes in this vulnerable young adult population. This study seeks to refine the YORS intervention through stakeholder input and pilot iterative testing followed by an efficacy randomized controlled trial. This project will significantly contribute to our knowledge base of practical strategies to address the opioid crisis.

DETAILED DESCRIPTION:
Young people are disproportionately affected by the current opioid crisis including worse retention and outcomes compared to older adults. Further, young adults typically do not have access to medications for opioid use disorder (OUD), and for those that do, struggles with adherence are a major barrier. Standard approaches to treatment typically do not incorporate developmentally informed strategies for engagement, retention, and medication adherence for this special population.

The Youth Opioid Recovery Support (YORS) model is an innovative wrap-around approach that attempts to address barriers to treatment engagement in this vulnerable young adult population, especially difficulties with medication adherence. Its components include: (1) Home delivery of extended release naltrexone (XR-NTX) for OUD; (2) Engagement of families in collaborative treatment planning and monitoring focusing on medication adherence; (3) Assertive outreach from the treatment team including actively tracking and communicating with youth and families by text messaging and social media to promote engagement and adherence; and (4) Contingency management to provide incentives for medication adherence. YORS is currently showing very promising results in a small pilot randomized clinical trial (RCT) by the investigative team.

The investigators propose to refine and then conduct a more definitive test of the YORS intervention for youth with OUD. In the first phase the investigators will conduct stakeholder focus groups to get input and feedback on potential refinements, while also conducting 3 cycles of pilot testing of these potential refinements. Based on the preparation and final synthesis of the intervention refinements, in the second phase the investigators will conduct an RCT to test the efficacy of YORS, by randomizing N=120 young adults ages 18-26 seeking treatment for OUD with XR-NTX at Mountain Manor Treatment Center (MMTC), to either the refined YORS intervention or treatment as usual (TAU) for a 6-month course of treatment with XR-NTX.

The primary outcome will be number of XR-NTX doses received. Secondary outcomes will include opioid relapse, days of opioid use, time to first opioid relapse, HIV risk behaviors, criminal behaviors, psychiatric symptoms, and family member distress and self-efficacy. It is hypothesized that participants in the YORS condition will receive significantly more XR-NTX doses and will demonstrate less severe opioid use and associated behaviors compared to those in the TAU group. The assertive YORS intervention has the potential to improve the real-world effectiveness and public health impact of medication for OUD in this very high-risk, vulnerable population. If the refined YORS intervention is found to be efficacious, it would set the stage for future work including: an economic analysis, a larger multi-site study, longer intervention duration, study of extended release buprenorphine, and study of step-down to less intensive interventions.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-28
* OUD diagnosis
* Willing (intending) to receive treatment with XR-NTX or XR-BUP under the care of a MTC physician/nurse practitioner
* Willingness to designate family member (or other suitable treatment significant other) for treatment involvement (i.e., a treatment significant other; TSO)

Exclusion Criteria:

* Psychiatric or medical instability (e.g., suicidality, psychosis, Sickle Cell disease with frequent crises) that would preclude participation in the trial
* Living situation (location greater than 75 miles from the center, homelessness) that would preclude participation in the trial

Ages: 18 Years to 28 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2020-02-17 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Number of MOUD injections received (XR-NTX or XR-BUP) | Treatment week 0 to 26 weeks
  Total number of injections received within 26 weeks
Rate of opioid relapse during the study period | Time Frame: Data measured every 2 weeks for the duration of the 26-week study period
  Relapse = 10 days of use within a 28 day period. Days of opioid use will be assessed through urine toxicology and self report methods.

CONTACTS AND LOCATIONS:
Overall Officials: Marc Fishman, MD, Principal Investigator — Maryland Treatment Centers
Locations (1):
- Mountain Manor Treatment Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No